CLINICAL TRIAL: NCT07032857
Title: Breaking Barriers: A Clinical Experimental Study of Intestinal Permeability in Children With Autism Spectrum Disorder
Brief Title: Intestinal Permeability in Children With Autism Spectrum Disorder
Acronym: IP-ASD
Status: Recruiting | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Prof, University of Bari
Other Study IDs: IP-ASD
Record Dates: First submitted 2025-06-10; First posted 2025-06-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorders
Keywords: autism spectrum Disorders; Intestinal permeability; Leaky gut
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 24hr Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism spectrum disorders: Intestinal Permeability Assessment
- Sibilings: Intestinal Permenability Assessmnt

SUMMARY:
In recent years, increasing attention has been directed toward the role of the gut-brain axis in the pathogenesis of neurodevelopmental disorders, particularly Autism Spectrum Disorder (ASD). Among the multiple contributing factors, the integrity of the intestinal barrier appears to play a crucial role. Enhanced paracellular permeability ("leaky gut") may allow luminal antigens and microbial metabolites to translocate into the systemic circulation, triggering inflammatory responses that could impact neuropsychological functioning.

Several studies suggest that, although intestinal permeability is not universally altered in all individuals with ASD, there exists a subset characterized by selective epithelial dysfunction, especially associated with repetitive and stereotyped behaviors.

This project aims to investigate, through a controlled sibling-based design, whether intestinal permeability indices are significantly altered in children with ASD and whether such alterations are specifically correlated with behavioral domains assessed through the ADOS instrument.

DETAILED DESCRIPTION:
Study Objectives

Primary Objective:

• To compare intestinal permeability profiles in children with ASD and their neurotypical siblings, using the La/Ma ratio and the recovery of specific sugars (lactulose, mannitol, sucrose, sucralose).

Secondary Objectives:

* To explore the correlations between intestinal permeability markers and behavioral dimensions assessed via ADOS, with particular focus on stereotyped behaviors and communication.
* To assess the presence of intestinal inflammation through fecal calprotectin (FC) measurement.

Study Design Observational, case-control, single-center clinical study involving children with ASD and unaffected siblings. The intra-family design allows for control of shared environmental and genetic factors.

Study Population

ASD Group (cases):

* Children with a clinical diagnosis of ASD according to DSM-IV, confirmed by ADOS-G.
* Aged between 2 and 14 years.

Control Group (siblings):

* Unaffected siblings who underwent expert clinical evaluation to exclude neurodevelopmental disorders.
* SCQ score below the risk threshold for ASD.

Experimental Methodology 7.1 Intestinal Permeability Test (IPT)

* Fasting and abstention from NSAIDs/alcohol for at least 72 hours.
* Baseline urine sample collection.
* Oral administration of a sugar cocktail containing:

  * Lactulose 5 g
  * Mannitol 1 g
  * Sucrose 20 g
  * Sucralose 1 g
* Collection of all urine passed during the following 6 hours.
* Samples stored at -80°C with sodium azide.

Biochemical Analyses

* Sugar quantification via UPLC-MS/MS (Waters ACQUITY™).
* Use of isotopically labeled internal standards and seven-point calibration curves.
* Calculation of urinary recovery percentages and La/Ma ratio.
* FC measured via ELISA (Calprest®). Behavioral Assessment Tools
* ADOS-G: severity assessment in communication, social interaction, and stereotyped behavior domains.
* SCQ: ASD screening in controls.
* IQ assessed with standardized psychometric tests.

Statistical Analysis

* Descriptive statistics using mean ± SD or median (IQR).
* Shapiro-Wilk test for normality.
* Welch's t-test or Mann-Whitney U test for group comparisons.
* Fisher's exact test for categorical variables.
* Spearman's rank correlation (ρ) for associations between permeability indices and behavioral variables.

Relevance and Future Perspectives This protocol contributes to the growing body of translational research exploring the impact of intestinal function on neurodevelopmental disorders. The potential to identify biomarkers associated with specific behavioral domains may inform future personalized therapeutic strategies, including those targeting the intestinal barrier through prebiotics, probiotics, or anti-inflammatory nutraceuticals.

ELIGIBILITY:
* Children with a clinical diagnosis of ASD according to DSM-IV, confirmed by ADOS-G.
* Consumption of a gluten-containing diet.
* Negative celiac disease serology (EMA and anti-TG2 IgA antibodies).
* Absence of IgE- or non-IgE-mediated food allergies.

Exclusion Criteria:

* Known neurological disorders.
* Major congenital anomalies.
* Severe head trauma.
* Chronic gastrointestinal diseases.
* Special diets (e.g., gluten-free or gluten/casein-free).
* Antibiotic or probiotic/prebiotic intake in the previous 4 weeks.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with a clinical diagnosis of ASD according to DSM-IV, confirmed by ADOS-G.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
intestinal permeability | baseline
  La/Ma ratio and the recovery of specific sugars (lactulose, mannitol, sucrose, sucralose).

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Bari Aldo Moro, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided